CLINICAL TRIAL: NCT03614390
Title: Mindfulness for Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Clinical assistant professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUHK-mind
Record Dates: First submitted 2018-07-31; First posted 2018-08-03 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Mindfulness; Burnout, Professional
MeSH Terms: conditions — Burnout, Professional | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBCT group (Other): There is only 1 arm in the study.
  The MBCT will be conducted according to the treatment manual. The program consists of eight weekly sessions. In between sessions, participants are advised to practice mindfulness meditations for 40-50 minutes every day.
  The teachers of the program will teach on voluntary basis. The teachers must have attended the 1-year foundation course to teach mindfulness (available in the United Kingdom and Hong Kong), regular mindfulness practice and must have at least yearly mindfulness retreat. This is in accordance to the good practice guidelines developed in the UK for mindfulness teachers
  Interventions: Behavioral: mindfulness based cognitive therapy (MBCT)

INTERVENTIONS:
Behavioral: mindfulness based cognitive therapy (MBCT) — a well described and structured intervention, which is published previously. The psychoeducation materials in the MBCT will be titrated to discuss about low mood and burnout

SUMMARY:
Burnout is common among medical students. Previous studies had shown that mindfulness based interventions may improve burnout and quality of life in medical students. Mindfulness-based cognitive therapy (MBCT) is one of the most often used mindfulness based interventions.

Medical students in the Chinese University of Hong Kong are invited to a MBCT on voluntary basis. They will be asked to fill in questionnaire that measures burnout, depression/anxiety, quality of life, and mindfulness at beginning and end of the MBCT. The pre-group and post-group data will be compared and analysed

ELIGIBILITY:
Inclusion Criteria:

* Medical students studying in Chinese University of Hong Kong

Exclusion Criteria:

* The investigators did not set any exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Maslach Burnout Inventory (MBI) | 8 weeks (before and after MBCT; after 8 weekly sessions)
  The validated Maslach Burnout Inventory (MBI) is a 22-item questionnaire that assesses three aspects of professional burnout syndrome which includes emotional exhaustion, depersonalization and lack of personal accomplishment. It is widely used in research and has been widely used in studies about medical student well-being. In the scale, burnout is conceptualized as a continuous construct and participant is asked to rate their job related feelings using a 7-point Likert scale ranging from "never" to "everyday". A high degree of burnout is defined as a respondent who scores low on the Personal Accomplishment subscale but high in the Emotional Exhaustion and Depersonalization subscales of the instrument

SECONDARY OUTCOMES:
21-item Depression Anxiety Stress Scale (DASS-21) | 8 weeks (before and after MBCT; after 8 weekly sessions)
  The 21-item DASS-21 questionnaire will be used to assess the presence of depression, anxiety and tension/stress with 7 items per subscale. Each item is ranked from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). The total score is computed by adding scores of each item and multiplying them by a factor of 2. Therefore, the total possible score ranges from 0 to 126. The questionnaire exhibits adequate validity and internal consistency among clinical and non-clinical samples
the World Health Organization Quality of Life Assessment (WHOQOL-BREF) | 8 weeks (before and after MBCT; after 8 weekly sessions)
  The WHOQOL-BREF consisted of 26 items representing four underlying domains: environment, psychological, social relationship and physical health. Scores within each domain can be transformed to a scale of 0-100, with higher scores represent better quality of life. The scales was used in medical students' burnout research
Five Facet Mindfulness Questionnaire (FFMQ) | 8 weeks (before and after MBCT; after 8 weekly sessions)
  The FFMQ consisted of 39 items representing five underlying constructs: observing, describing, acting with awareness, non-judging of inner experience and non-reactivity to inner experience. Each item is rated from 1 ("never or very rarely true) to 5 ("very often or always true"). Total Score can be obtained by summation of scores.The higher score represents a more mindful attitude in daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- Lek Yuen Clinic, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available on request from other researchers